CLINICAL TRIAL: NCT04946695
Title: Feasibility and Efficacy of the Use of Telephysiotherapy for Improving Functional Independence and Quality of Life in Children and Young People With Lower Limb Fracture in a Low Resource Setting in Anantapur (India)
Brief Title: Feasibility and Efficacy of the Use of Telephysiotherapy in Anantapur
Acronym: Telefisio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Maria Jose Estebanez Perez, Feasibility and Efficacy of the Use of Telephysiotherapy in Anantapur, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15031973
Record Dates: First submitted 2021-06-10; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Lower Extremity Fracture
Keywords: telephysiotherapy; fracture; low resources; paediatrics
MeSH Terms: conditions — Fractures, Bone | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: This research is a quasi-experimental multicentre pre-post intervention pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telefisio India (Experimental): Feasibility and efficacy of the use of Telephysiotherapy for improving functional independence and quality of life in children and young people with lower limb fracture in a low resource setting in Anantapur (India).
  Interventions: Other: Telefisio India

INTERVENTIONS:
Other: Telefisio India — Implement telephysiotherapy programmes in low-resource areas.
  Other Names: Improving functional independence and quality of life in low-income areas

SUMMARY:
Injuries remain the most frequent cause of mortality in children and young people. Studies with: telephysiotherapy programmes have published results of effectiveness, validity, non-inferiority and important advantages, providing an opportunity to define new health and social intervention policies.

In rural regions such as Anantapur, there are few physiotherapists compared to the potential need; innovative strategies are needed to improve access to more specialised physiotherapy care. There is also a significant paucity of studies in low resources geographies, making this research highly justified.

This research is a quasi-experimental multicentre pre-post intervention pilot study in a population aged 5-16 years with a diagnosis of lower limb fracture in Anantapur (India).

The main objective is to assess the feasibility and efficacy of using a 4-week personalised telephone therapy programme, as well as adherence, identify barriers to use and satisfaction with the intervention.

Subjects will receive a baseline assessment (T0-pre) obtaining data on Physical Function (TUG), Functional Independence (FIM), Activities of Daily Living (ADL) and Quality of Life (ISF-12). At the end of the intervention (T1-post) a new evaluation of the outcome variables will be carried out by adding data on adherence, barriers to use and satisfaction (ad hoc questionnaire and TSQ).

This research should provide insights into the possibility of implementing telephone therapy programmes in hospital settings in low resources areas.

DETAILED DESCRIPTION:
This research is a quasi-experimental multicentre pre-post intervention pilot study in a population aged 5-16 years with a diagnosis of lower limb fracture in Anantapur (India).For the development of this research a non-probabilistic purposive sampling will be used for the convenience of the study, n=30

The main objective is to assess the feasibility and efficacy of using a personalised telephysiotherapy programme for improving functional independence and quality of life in children and young people with lower limb fracture in a low resource setting in Anantapur.

Secondary objectives:- To assess the frequency and distribution of injuries among study subjects.- To evaluate the satisfaction with the telephysiotherapy programme in rural areas with low resources of the participants. - To analyze the degree of adherence to the telephysiotherapy treatment.- To identify obstacles and possible barriers in the development of the intervention.

Participants in the study will receive a personalised telephysiotherapy programme adapted to their injury for 4 weeks.

For the monitoring of the telephysiotherapy programme, the participants will receive a free recycled mobile device.

This device, as well as their intervention programme ,designed thanks to the Physiotec software , will be updated weekly by the research team and the hospital physiotherapist.

The personalised programme describes the exercises to be performed, the number of sets and repetitions and the progression criteria, which will be based on published clinical guidelines for patients with lower limb fractures.

Participants and their relatives will be instructed to perform the self-training by following the exercises on video through the programme to be carried out.

The investigators will consider three types of outcomes for this research study:

- Affiliation data and demographic outcomes: Name and surname, Contact Details, Age variable and Gender variable

- Primary explanatory outcomes: Physical Function, (TUG test), Functional Independence (FIM scale), , Activities of Daily Living variables (IB) and quality of life(SF-12 questionnaire)

- Secondary explanatory outcomes.Type of injury variable ,Adherence to treatment variable , and Variable Satisfaction, Obstacles and Barriers to the use of tele-physiotherapy (ad hoc questionnaire and TSQ).

Data collection will be carried out:

T0-pre intervention :

Physical Function (TUG), Functional Independence (FIM), Activities of Daily Living (IB) and Quality of Life (SF-12). Type of injury (medical history).

T1-post intervention:

A new evaluation of the outcome variables will be carried out by adding data on barriers to use and satisfaction (ad hoc questionnaire and TSQ).

Weekly check-ups :

Adherence to treatment will be measured by the application and during by the medical service.

The fundamental ethical precepts according to the Declaration of Helsinki and Law 14/2007 of 3 July on Biomedical Research will be respected, guaranteeing the protection and confidentiality of the data in accordance with the provisions of Organic Law 3/2018, of 5 December,, on the Protection of Personal Data (LOPD).

In order to carry out the study, acceptance will be requested from the Research Ethics Committee.

A document has been drawn up that includes the Informed Consent and prior information about the research, which must be signed by the legal guardians of the participants in the study.

Be informed of the possibility to revoke the consent given at any time, without having to justify its decision and without prejudice.

This research should provide knowledge on the possibility of implementing tele-physiotherapy programmes in a low resource setting.

The possible limitations:

Misuse of devices ,Technical problems, Lack of Internet connectivity,... The appearance of selection and information biases The possible alteration of the relationship dynamic between patients and their relatives and the medical team.

Lack of improvement and positive evolution of the patient Difficulty in obtaining the necessary resources.

In conclusion, the positive results of this intervention mean that the investigators are looking at an improvement in accessibility to specialised health care, an improvement in the quality of care received and a reduction in health care costs in terms of hospital admissions, health Centre care and travel for the health care needed today in Anantapur (India).

Thank you

ELIGIBILITY:
Inclusion Criteria:

* Children (aged 5-16 years) living in rural areas with referral hospitals Bathalapali and Kaliandur.
* Diagnosed by the medical team of these hospitals with lower limb fracture.
* Children and/or responsible family members must have reading and writing skills in English or Telugu (language of the Anantapur region).

Exclusion Criteria:

- Presence of a diagnosis of neurological, mental or infectious disease, cognitive disorder and/or comorbidities to musculoskeletal involvement.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The Barthel Index (Functional Independence) | Four weeks
  Independence in self-care and mobility; it assesses the patient's level of independence with respect to the performance of some basic activities of daily living (ADLs), whereby different scores are assigned. Provides information both from the global score and from each of the partial scores for each activity. This helps to gain a better understanding of the person's specific impairments and facilitates the assessment of their evolution over time. The total score is reached by adding up the scores for each measurement and predicts the time and help that the patient will require. Scores can range from zero to 100, adding up to five points per category, so that higher scores indicate a greater degree of functional independence. It is an easy to apply measure, with a high degree of reliability and validity, capable of detecting changes, easy to interpret, and is not bothersome to apply.
The functional independence measure (FIM) | Four weeks
  A global ordinal scale for functional assessment (mobility and self-care) is useful in making decisions about the effectiveness of therapy. Several studies have used the FIM to investigate treatment outcome in self-care, transfers (mobility) and locomotion. The FIM uses a 7-level scale to rate functional performance. The total FIM score is obtained by summing the ratings of the 18 items included in the different levels. The scale has good reliability and its comparison with other instruments yields correlations of 0.84 with the Barthel Index.
The Timed "Up & Go" test (TUG) Functional mobility | Four weeks
  The original Get-up and Go test was intended to clinically assess dynamic balance in older people during the performance of a task involving fall-critical situations. The TUG test measures, in seconds, the time required for an individual to get up from a standard chair with armrests (approximately 46 cm high), walk 3 m, turn around, return to the chair and sit down again. The test has been widely used in clinical practice as an outcome measure to assess functional mobility, fall risk or dynamic balance in adults. The TUG test, proved to be a good tool for assessing functional mobility in the paediatric. Assessment in seconds, ranging from less than 10 seconds considered as independent mobility to more than 20 seconds considered as reduced mobility.
Quality of life (SF12), 12- Item Short Form Survey | Four weeks
  The SF-12 questionnaire will be used for the assessment of health-related quality of life. The SF-12 questionnaire assesses eight dimensions of health-related quality of life: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. The range of scores obtained is from 0 to 63 points. High internal consistency indices are observed both in the Spanish validation of the questionnaire 0.83 and 0.9039, as well as in several international studies.

SECONDARY OUTCOMES:
Adherence to treatment | Four weeks
  The telephone therapy application automatically records compliance with the scheduled sessions, as well as the non-compliance with the protocol indicated by the physiotherapist. This adherence is completed by the weekly control with the physiotherapist at the reference hospital, who will record attendance at the sessions.
Satisfaction, Obstacles and Barriers to the use of tele-physiotherapy, Satisfaction ad hoc questionaire | Four weeks
  The investigators will use a questionnaire designed Ad hoc which includes a Likert scale (1 Dissatisfied - 5 Very satisfied), and open questions for the patient and relatives to point out the possible obstacles and barriers in the use of TelePhysiotherapy.
Satisfaction, Obstacles and Barriers to the use of tele-physiotherapy, TSQ (Telemedicine Satisfaction Questionnaire) | Four weeks
  The TSQ is a 14-item questionnaire in its final version, the questionnaire items are scored on a five-point scale, from 1 being strongly disagree to 5 being strongly agree.. The internal consistency of the TSQ was 0.93, which is considered acceptable and indicates strong correlations between the items that make up the scale. Predictive validity supported the conclusion that the TSQ measured patient satisfaction with telemedicine (Pearson's correlation coefficient (r=0.45, P<0.05) (36).
% of patients with type of injury | Pre-intervention
  The investigators will estimate this as a nominal qualitative variable; this variable coincides with the diagnosis provided by their doctor in one of the reference hospitals.

OTHER OUTCOMES:
First name and surname: | Pre-intervention
  The investigators will estimate it with a research identification code as a numeric variable (e.g. Id-001).
Contact Details | Pre-intervention
  The investigators will identify it as a Nominal qualitative variable.
Age | Pre-intervention
  Age will be estimated as a numerical variable.
Gender | Pre-intervention
  Gender will be identified as a nominal categorical variable, indicating whether it is Male or Female, coded with "1" and "2", respectively.

CONTACTS AND LOCATIONS:
Overall Officials: María Jose MJ Estebanez- Pérez, MSC, PT, Principal Investigator — University of Málaga (Spain)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estebanez-Perez MJ, Martin-Valero R, Moreno-Morales N, Linan-Gonzalez A, Fernandez-Navarro R, Pastora-Bernal JM. Digital physiotherapy intervention in children in a low resource setting in Anantapur (India): Study protocol for a randomized controlled trial. Front Public Health. 2022 Sep 30;10:1012369. doi: 10.3389/fpubh.2022.1012369. eCollection 2022. PMID 36249182